CLINICAL TRIAL: NCT00885976
Title: The Predictors and Patient Versus Parental Perceptions of Health-Related Quality of Life in Pediatric Chronic Pain
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Thomas R. Vetter, MD, MPH, M.D., M.P.H., University of Alabama at Birmingham
Other Study IDs: F081114005
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Pediatric Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is intended to provide additional insight into the factors affecting health-related quality of life with pediatric chronic pain as perceived by the patient versus his or her parents.In doing so, additional insight into the subjective interpretation the pediatric chronic pain experience will be gained. The four objectives of this study will be (a) to examine further the relationship between patient self-reported health-related quality of life and parent proxy-reported health-related quality; (b) to identify what biological, psychological, and/or social factors are the strongest predictors of a pediatric chronic pain patient's self-reported pain intensity and self-reported health-related quality of life, in a diverse cohort of patients referred to and subsequently treated by an anesthesiology-based yet interdisciplinary pediatric chronic pain medicine program; (c) to assess the effect of patient-specific, pain-focused biopsychosocial treatment regimen on pain intensity and health-related quality of life; and (d) to determine the effect of patient/parental satisfaction with on-going health care on their compliance with and uptake of the pain treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* outpatients ranging between 8 years and 18 years of age directly referral from either their primary care physician or another specialist physician

Exclusion Criteria:

* patients in whose biologic families English is not the primary, native language
* patients suffering from severe cognitive dysfunction (i.e., mental retardation)
* patients with a life-expectancy of less than three months at the time of initial clinical evaluation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will come from those patients evaluated and treated in the Pediatric Chronic Pain Medicine Clinic at the Children's Hospital facilities. The likely study population includes essentially the pediatric population of the entire state of Alabama and immediately adjacent states (i.e., the geographic catchment area of the Children's Hospital of Alabama).
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Heath-related quality of life | Baseline at time of initial outpatient clinic visit
  PedsQLTM 4.0 and 36-Item Short-Form Health Survey Version 2 (SF-36v2)
Pain intensity and functional disability | Baseline at the time of initial outpatient clinic visit
  Pediatric Pain Questionnaire (PPQ) and Functional Disability Inventory (FDI)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Vetter, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Pediatric Chronic Pain Medicine Program at Children's Hospital, Birmingham, Alabama, United States

REFERENCES:
- [Result] Vetter TR, Bridgewater CL, McGwin G Jr. An observational study of patient versus parental perceptions of health-related quality of life in children and adolescents with a chronic pain condition: who should the clinician believe? Health Qual Life Outcomes. 2012 Jul 23;10:85. doi: 10.1186/1477-7525-10-85. PMID 22824550